CLINICAL TRIAL: NCT05543889
Title: Evaluation of Clinical Decisions and Assessment of Those at Risk of Primary Angle Closure by Community Optometrists
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: JINA1001
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-12

CONDITIONS: Angle Closure Glaucoma
Keywords: Limbal anterior chamber depth; Optometrist; Angle-closure; Van Herick
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 100 patient participants will be recruited for limbal anterior chamber depth image capture. These images will be used to develop the clinical vignette database
- Optometrists: 50 optometrists will be recruited to undertake the clinical vignette assessment
  Interventions: Other: Educational package

INTERVENTIONS:
Other: Educational package — Online learning package that will discuss the van Herick technique, grading, accuracy and information and discusses the current guidelines for primary angle closure suspect referral.
  Groups: Optometrists

SUMMARY:
Increases in the aging population has resulted in increased demand for glaucoma services. Glaucoma is a disease that if untreated, can lead to blindness. This increase and need for long term treatment with monitoring have resulted in a significant demand in the hospital eye service (HES). Many departments are now facing a considerable backlog of outpatient appointments and it's essential that these appointments are reserved for patients who are at risk of glaucoma blindness.

Primary angle closure (PAC) glaucoma is a type of glaucoma, where the drainage route for the fluid inside the eye (known as the angle) is narrowed or blocked. It has been recently identified that approximately half of patients referred into the HES for a suspect narrow angle for further investigation are healthy and are immediately discharged. The exact reasons for these findings are unknown.

This project will investigate clinical decisions by community optometrists who account for the majority of PAC referrals into the HES, as well as assessing their ability to evaluate those at risk of PAC. This project will also examine whether clinical agreement could be improved by providing an educational package.

A clinical image database of angles will be acquired from glaucoma patients attending Moorfields Eye Hospital. A learning package discussing angle closure referral will also be developed. Community optometrists will be invited to complete a questionnaire on their clinical decision making. This will be followed by the vignette assessment, learning package and re-assessment.

If this educational package and/or any other identifiers are found to improve agreement levels, this could reduce the number of referrals and enable community monitoring of those at low risk of developing PAC glaucoma in their lifetime.

ELIGIBILITY:
Inclusion Criteria:

New patients attending the glaucoma clinic at Moorfields Eye Hospital

Exclusion Criteria:

* They cannot be examined using a table mounted slit lamp due to physical limitations or have gross nystagmus.
* Unable to consent
* If they are unable to communicate in English and there is no available interpreter that meets requirements set out by Moorfields standard operating policies for patients
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New patients to the glaucoma service will be selected as they would be a real-world reflection of those who have been identified at risk of developing glaucoma that have been referred for glaucoma investigation within the hospital eye service from primary care. Furthermore, they would have an enriched sample of narrow angles that are required to achieve the desired the case-mix required for the image database within the set timelines.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-03-07 (Estimated); Study Completion 2024-03-07 (Estimated)

PRIMARY OUTCOMES:
Agreement of community optometrists on measuring Limbal anterior chamber depth | 12 months
  Levels of agreement and precision of optometrist observers before and after intervention of online educational package in assessment of Limbal anterior chamber depth as a surrogate measure of angle width. Agreement will be measured via an online assessment vignette assessment package. Weighted Kappa statistic and levels agreement will be the outcome measures

SECONDARY OUTCOMES:
Qualitative outcome measures from optometrists | 12 months
  Questionnaire based outcomes capturing data around current practice, qualifications and training, knowledge and resources available in practice with regards to angle closure diagnosis and referral
Qualitative outcome measures from patients | 12 months
  Difficulty in performing tests and satisfaction from the appointment (Likert scale 1-10), time taken (minutes) and costs of travel (£) to test site and waiting time to be examined from referral (months).

CONTACTS AND LOCATIONS:
Overall Officials: Anish Jindal, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust/UCL
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No